CLINICAL TRIAL: NCT05168371
Title: Pilot RCT for Cognitive-Behavioural & Mindfulness-Based Online Programs for Female Sexual Dysfunction
Brief Title: Cognitive-Behavioural & Mindfulness-Based Online Programs for Female Sexual Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-03914
Record Dates: First submitted 2021-11-23; First posted 2021-12-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Female Sexual Dysfunction
Keywords: Sexual Desire; Mindfulness; Cognitive Behavioral Therapy; Cognitive Behavioural Therapy; Mindfulness Based Therapy; Digital Health; Sexual Interest/Arousal Disorder; Female Sexual Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-O (Experimental): Women randomized to this arm will receive access to the eight modules of Cognitive-Behavioural Therapy-Online (CBT-O). Participants will meet weekly via Zoom with treatment navigators during the 8-12 weeks that it takes to complete the program.
  Interventions: Behavioral: Cognitive-Behavioural Therapy - Online (CBT-O)
- MBT-O (Experimental): Women randomized to this arm will receive access to the eight modules of Mindfulness-Based Therapy-Online (MBT-O). Participants will meet weekly via Zoom with treatment navigators during the 8-12 weeks that it takes to complete the program.
  Interventions: Behavioral: Mindfulness-Based Therapy - Online (MBT-O)
- Wait-List Control (No Intervention): Participants who are randomized to the wait-list group will complete two baseline online questionnaire/assessment batteries before being randomized to one of the active treatment groups. Participants will be randomized into one of the active treatment groups after a 10 week waiting period.

INTERVENTIONS:
Behavioral: Cognitive-Behavioural Therapy - Online (CBT-O) — Face-to-face CBT was adapted for web-based self-directed therapy. CBT-O was found to be feasible and usable (Stephenson et al., 2021; Zippan et al., 2020).
  Each of the eight modules has between-module activities to complete. The eight modules are: 1) Psychoeducation, introduction to CBT; 2) The cognitive model and thought records; 3) Unhelpful thinking patterns; 4) Cognitive restructuring; 5) Behavioral experiments; 6) Self-touch and sensate focus; 7) Sensate focus with your partner; and 8) Maintaining (and extending) your gains.
  Arms: CBT-O
Behavioral: Mindfulness-Based Therapy - Online (MBT-O) — The content of MBT-O was adapted from an efficacious face-to-face mindfulness intervention for women with Sexual Interest/Arousal Disorder (Brotto et al., 2021; Paterson et al., 2017). MBT-O was found to be feasible and usable (Brotto et al., under review).
  Each of the eight modules has between-module activities to complete. The eight modules are: 1) Psychoeducation, introduction to mindfulness; 2) Increasing awareness of physical sensations in the body; 3) Exploring movement and body image; 4) Awareness of sexual thoughts and beliefs; 5) Working with aversion, self-touch; 6) Exploring sexual sensations, knowing limits; 7) Integrating the partner into mindful touching; and 8) Maintaining (and extending) your gains.
  Arms: MBT-O

SUMMARY:
Female sexual dysfunction (FSD) affects approximately one-third of women worldwide and is linked to negative physical, psychological, and interpersonal outcomes. Although both cognitive-behavioral therapy and mindfulness-based therapy are effective treatments for FSD, face-to-face treatments can be costly and are inaccessible to many people in remote areas. The goal of the current study is to pilot a randomized controlled trial to examine the effectiveness of and satisfaction with two online interventions for FSD. Women will be randomized to an online cognitive-behavioral program, an online mindfulness-based program, or a wait-list control group. Treatment will be administered entirely online and last 8-12 weeks. Women will meet weekly via Zoom with a navigator who will provide individualized support.

DETAILED DESCRIPTION:
HYPOTHESES:

1. Compared to women in the wait-list control arm, women in the CBT and MBT arms will have significant post-treatment and follow-up improvements in self-report measures of the primary outcomes: (a) sexual distress and (b) sexual desire.
2. Compared to women in the wait-list control arm, women in the CBT and MBT arms will have significant post-treatment and follow-up improvements in self-report measures of the secondary outcomes: (a) overall sexual function, (b) sexual satisfaction, (c) relational sexual concern, (d) satisfaction with life, and (e) relationship satisfaction.
3. Improvements in depression, sexual avoidance, and sexual consequences will significantly mediate improvements in primary outcomes at all post-treatment assessment points.
4. Higher levels of baseline relationship satisfaction, higher levels of partner involvement, more positive baseline expectations about treatment efficacy, higher levels of treatment compliance, and perceiving higher levels of empathy and effectiveness from navigators will predict greater improvements in primary outcomes at post-treatment and follow-up.
5. Baseline personality will moderate intervention effects at post-treatment and follow-up.
6. Women in both the CBT and MBT arms will report being satisfied with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cis and trans women of any sexual orientation.
* Must be fluent in English (online materials delivered in English).
* Must have consistent access to the internet, basic competency in using online platforms (self-report).
* Must be in a committed, stable romantic relationship of at least 6 months (because aspects of the interventions require partner participation). Partners may be of any gender.
* Must meet telephone screening diagnostic criteria for sexual interest/arousal disorder.
* Must be sexually active with a partner over the preceding 4 weeks (due to the sexual function outcome measure), and willing to engage in sexual activity with their partner during the study.
* Must be able to participate in an 8-12-week online treatment.

Exclusion Criteria:

* Have sexual dysfunction that is, in their estimation, fully attributable to another psychiatric diagnosis, the effect of a substance, a general medical condition (e.g., Multiple Sclerosis), or non-sexual conflict in the relationship, none of which are meant to be addressed by the proposed interventions.
* Poorly managed Anxiety or Mood Disorder (as per degree of life interference assessed at screening).
* Report visual impairments that would make it difficult to read online materials.
* Are regularly using prescription narcotics illegal recreational drug (not including cannabis).
* Plan to change their medications known to impact sexual function over the course of the study.
* On assessment report plans to end their romantic relationship in the next 6 months.
* Engage in any other treatment for their sexual difficulties during the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 129 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in sexual distress | baseline; mid-treatment (an average of 5 weeks after starting the 8-module program); post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  Revised version of the Female Sexual Distress Scale-R (Derogatis et al., 2008). Scores on the scale range from 0-52, where higher scores represent higher levels of distress.
Change in sexual desire | baseline; mid-treatment (an average of 5 weeks after starting the 8-module program); post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  The Sexual Interest and Desire Inventory (SIDI; Clayton et al. 2006) total score will be used to measure sexual desire. Possible total scores range from 0-51, with higher scores indicating higher levels of sexual functioning.

SECONDARY OUTCOMES:
Change in sexual function | baseline; mid-treatment (an average of 5 weeks after starting the 8-module program); post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  Female Sexual Function Index total score (FSFI; Rosen et al., 2000). Scores range from 2 - 36 where increase in sexual dysfunction is represented by lower scores.
Change in sexual satisfaction | baseline; post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  Quality of Sex Inventory (QSI; Shaw & Rogge, 2016). For all items, responses are given values on a 0 to 5 point scale with 0 = Not at all TRUE and 5 = Completely TRUE. The items of the sexual satisfaction subscale are summed to create a total where higher scores indicate higher levels of sexual satisfaction (0-60). The items of the sexual dissatisfaction subscale are summed separately to create a total where higher scores reflect higher levels of sexual dissatisfaction (0-60).
Change in relational sexual concern | baseline; post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  Relational concern subscale of the Sexual Satisfaction Scale-Women (SSS-W; Meston & Trapnell, 2005). Scores range from 6-30, with higher scores reflecting lower levels of sexual relational concern.
Change in relationship satisfaction | baseline; post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  Couples satisfaction index (CSI-16; Funk & Rogge, 2007). CSI-16 scores can range from 0 to 81. Higher scores indicate higher levels of relationship satisfaction.
Treatment satisfaction for module 1 | An average of 1 week after starting the 8-module program
  Face-valid single item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing module 1.
Treatment satisfaction for module 2 | An average of 2 weeks after starting the 8-module program
  Face-valid single item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing module 2.
Treatment satisfaction for module 3 | An average of 3 weeks after starting the 8-module program
  Face-valid single item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing module 3.
Treatment satisfaction for module 4 | An average of 5 weeks after starting the 8-module program
  Face-valid single item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing module 4.
Treatment satisfaction for module 5 | An average of 6 weeks after starting the 8-module program
  Face-valid single item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing module 5.
Treatment satisfaction for module 6 | An average of 7 weeks after starting the 8-module program
  Face-valid single item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing module 6.
Treatment satisfaction for module 7 | An average of 9 weeks after starting the 8-module program
  Face-valid single item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing module 7.
Treatment satisfaction for module 8 | An average of 10 weeks after starting the 8-module program
  Face-valid single item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing module 8.
Quantitative program treatment satisfaction as assessed by the adapted Erectile Dysfunction Inventory of Treatment Satisfaction | post-treatment (within 2 weeks of completing the 8-module program)
  Adapted Erectile Dysfunction Inventory of Treatment Satisfaction (Althof et al., 1999; items 1-10). Scores range from 0-40, with higher scores reflecting higher treatment satisfaction.
Qualitative program treatment satisfaction | through completion of the 8-module program, an average of 10 weeks
  Qualitative feedback about eSense and between-module activities collected by treatment navigators.
Change in satisfaction with life | baseline; post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  Satisfaction with Life Scale (Diener et al., 1985). Scores range from 5-35, with higher scores reflecting higher levels of life satisfaction.

OTHER OUTCOMES:
Change in depression (mediator) | baseline; mid-treatment (an average of 5 weeks after starting the 8-module program); post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  Patient Health Questionnaire (PHQ-9). Scores can range from 0-27, with higher scores indicating more depression symptoms.
Change in sexual avoidance (mediator) | baseline; mid-treatment (an average of 5 weeks after starting the 8-module program); post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  The Golombok Rust Inventory of Sexual Satisfaction (GRISS) Questionnaire (female) - Sexual Avoidance Subscale. Scores can range from 0-16, with higher scores indicating higher levels of sexual avoidance.
Change in sexual consequences (mediator) | baseline; mid-treatment (an average of 5 weeks after starting the 8-module program); post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  Measure of Sexual Consequences (Stephenson et al., 2018). Scores can range from 11-55, with higher scores indicating more frequent negative sexual consequences.
Participants' baseline expectations about treatment efficacy assessed by two face-valid items (moderator) | baseline
  measured using two items: "To what extent to you think the treatment you will receive is logical in terms of alleviating your sexual desire concerns?" and "To what extent do you expect improvement in your sexual desire as a result of this treatment?"
Treatment compliance: Single-item measure of between-module activity completion (moderator) | through completion of the 8-module program, an average of 10 weeks
  navigators will ask participants to rate between-module activity completion on a 1-7 Likert scale ranging from "did not attempt" to "successfully completed all assignments" weekly
Treatment compliance: Between-module activity completion assessed by Homework Rating Scale-II (moderator) | through completion of the 8-module program, an average of 10 weeks
  participants complete the Homework Rating Scale-II (HRS-II) after each module. Scores can range from 0-48, with higher scores reflecting high levels of between-module activity completion.
Treatment compliance: Navigator adherence to study guidelines (moderator) | through completion of the 8-module program, an average of 10 weeks
  measuring navigator adherence to study guidelines by recording a random 50% of Zoom sessions (participants will be informed of these recordings) and coding navigator sessions for adherence using an adherence measure developed by investigators that access adherence to study guidelines, with higher scores reflecting higher levels of adherence to study guidelines.
Treatment compliance: Number of weeks in program (moderator) | post-treatment (within 2 weeks of completing the 8-module program)
  Recording number of weeks participant took to complete the program.
Treatment compliance: Number of treatment sections of program completed (moderator) | post-treatment (within 2 weeks of completing the 8-module program)
  Recording number of treatment sections participants complete.
Treatment compliance: Participant engagement with website as assessed by Google Analytics data (moderator) | through completion of the 8-module program, an average of 10 weeks
  eSense website engagement assessed by Google analytics data (e.g., total duration of time on website). This will provide a measure of participant engagement.
Perceived navigator empathy (moderator) | post-treatment (within 2 weeks of completing the 8-module program)
  Empathy subscale of the Barrett-Lennard Relationship Inventory (Barrett-Lennard, 2015). Scores range from -48 to 48, with higher scores reflecting that participants perceive higher levels of empathy in their navigator.
Perceived navigator alliance (moderator) | post-treatment (within 2 weeks of completing the 8-module program)
  Perceived navigator alliance with the Working Alliance Inventory, Short Form (Hatcher & Gillaspy, 2006). Scores range from 12-84, with higher levels reflecting that participants perceive higher levels of working alliance with their navigator.
Partner Involvement (moderator) | post-treatment (within 2 weeks of completing the 8-module program)
  Two face-valid questions asking how much their partners were involved with and supportive of their treatment. The items are: "How involved has your partner been with your participation over the course of your involvement with eSense (e.g., talking to you about your participation, viewing modules themselves, participating in activities)?" and "How supportive has your partner been of your participation in the eSense program?"
Big-Five personality traits (exploratory moderator) | baseline
  Big Five Inventory-10 (BFI-10; Rammstedt & John, 2007)
Change in PTSD symptoms (exploratory outcome) | baseline; mid-treatment (an average of 5 weeks after starting the 8-module program); post-treatment (within 2 weeks of completing the 8-module program); and 6-month follow-up
  PTSD Checklist (PCL) - 5; 4-item version (Price et al., 2016). Scores can range from 0-16, with higher scores indicating more severe PTSD symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Brotto, PhD, Principal Investigator — The University of British Columbia; Kyle Stephenson, PhD, Principal Investigator — Xavier University of Louisiana.
Locations (1):
- UBC Sexual Health Research Lab; Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Brotto LA, Stephenson KR, Marshall N, Balvan M, Okara Y, Mahar EA. Evaluating a Digital Health Tool Designed to Improve Low Sexual Desire in Women: Mixed-Methods Implementation Science Study. J Med Internet Res. 2025 Mar 25;27:e69828. doi: 10.2196/69828. PMID 40132194

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT05168371/Prot_SAP_001.pdf